CLINICAL TRIAL: NCT03097042
Title: Comparison of Two Different Catheter Withdrawal Technique During Embryo Transfer
Brief Title: Comparison of Two Different Catheter Withdrawal Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Çiğdem Yayla Abide, MD, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180/2016
Record Dates: First submitted 2017-01-24; First posted 2017-03-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Embryo; Catheter Site Discharge
MeSH Terms: interventions — Embryo Transfer

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): The catheter will be pulled back slowly and without rotation
  Interventions: Procedure: Embryo transfer with catheter Manipulation
- Control Group (Active Comparator): The catheter will be pulled back by rotating 360 degrees round itself
  Interventions: Procedure: Embryo transfer any further manipulation

INTERVENTIONS:
Procedure: Embryo transfer any further manipulation — The catheter will be pulled back slowly and without rotation with the plunger still pushed forward
  Arms: Control Group
Procedure: Embryo transfer with catheter Manipulation — catheter rotation during withdrawal
  Arms: Study group

SUMMARY:
The embryologist will oad the embryos into the catheter at the right position, then the catheter will be slowly pushed through the cervical canal, 1-2 cm beneath the fundus 5.5 cm away from the cervical external os.The embryos will be delivered by pushing the plunger of the syringe from the mid-cavitary positioned catheter and keeping the plunger pushed down.

Study Group: The catheter will be pulled back slowly and without rotation with the plunger still pushed forward.

Control Group: The catheter will be pulled back slowly with a 360°rotation with the plunger kept pushed forward.

DETAILED DESCRIPTION:
Patients to be included will be those meeting the study criteria who present at Istanbul Zeynep Kamil Training and Research Hospital, In vitro fertilization unit between February 1, 2017 and August, 2017.

The voluntary participants of the study will undergo controlled ovarian stimulation that is routinely performed in our clinic, followed by ovum pick up (OPU) and embryo transfer procedure. Volunteers will be asked to hold the urine 2 hours before the procedure to ensure fullness of the bladder. Identification details will be checked to verify that the names on the embryo containers are correct. The embryos will be examined by the embryologist. The participants will be informed before the procedure about the fertilization rates, number and quality of the developed embryos, the number of embryos to be transferred and the number of embryos planned to be frozen. Patients will undergo the procedure in the lithotomy position.The fullness of the bladder will be verified by inserting a speculum cervix and the vagina will be cleaned with a sterile serum physiological saline solution (SF) sponge, and cervical mucus aspired from the external os gently with a special soft aspirator catheter.

After the cervix is cleaned with culture liquid, a trial transfer will be performed with a sterile catheter. At this stage, only the soft internal catheter will pass through the internal os and the outer sheath will be stopped when it reaches the internal os. The outer sheath of the catheter will be advanced 2 cm into the cervical canal under ultrasound guidance and will be stopped before passing the internal os. Once it is ensured that the soft catheter is inside the endometrial cavity, the embryologist will be informed of the appropriate catheter position. Embryologist will oad the embryos into the catheter at the right position, then the catheter will be slowly pushed through the cervical canal, 1-2 cm beneath the fundus 5.5 cm away from the cervical external os. The embryos will be delivered by pushing the plunger of the syringe from the mid-cavitary positioned catheter and keeping the plunger pushed down. Afterwards, the volunteers will be randomly divided into two groups. Randomization will be ensured by a computer-based programme.

* 1st Group Volunteers: The catheter will be pulled back slowly and without rotation with the plunger still pushed forward.
* 2nd GroupVolunteers:The catheter will be pulled back slowly with a 360° rotation with the plunger kept pushed forward. The speculum will remain in the cervix until the embryologist checks the catheter for the presence of any embryos, blood or mucus.

Parameters to be Reviewed: Age, weight, height of the participants, primary/secondary infertility, infertility duration, presence of additional diseases, gravida, parity, abortion history, endometrial thickness on the day of HCG, infertility reasons, baseline and total gonadotropin dose, stimulation period, number of collected oocytes, number of M2 oocytes, quality of transferred embryos, BhCG positivity

ELIGIBILITY:
Inclusion Criteria:

Volunteers between the ages 20 to 40 Good quality embryo transfer Easy embryo transfer (use of soft catheter, not using tenaculum), Fresh cycle Single embryo transfer

Exclusion Criteria:

Volunteers younger than 20 and older than 40 years old Volunteers with poor ovarian reserve Low quality embryos Difficult embryo transfer (use of rigid catheter, use of tenaculum, passing of outer catheters heath from cervical os) Frozen cycle Volunteers that receive another transfer of embryos that remain in the catheter after the initial transfer.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy | 6 months
  Detection of the fetal heart rate by ultrasonography

SECONDARY OUTCOMES:
mucus or blood stained catheter | 6 months
  The rates of mucus and/or blood stained catheter will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Yayla Abide C, Ozkaya E, Sanverdi I, Bostanci Ergen E, Kurek Eken M, Devranoglu B, Bilgic BE, Kilicci C, Kayatas Eser S. Prospective Randomized Trial Comparing Embryo Transfers of Cases with and without Catheter Rotation during Its Withdrawal. Gynecol Obstet Invest. 2018;83(4):397-403. doi: 10.1159/000489493. Epub 2018 May 14. PMID 29758560